CLINICAL TRIAL: NCT02042872
Title: The Efficacy of Zoledronic Acid in the Prevention of Bone Loss in Acute Spinal Cord Injury
Brief Title: Zoledronic Acid Administration in Acute Spinal Cord Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Principal Investigator, William A. Bauman, M.D., Director VA RR&D Center of Excellence for the Medical Consequences of SCI, James J. Peters Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5481-03-0013; R-454-03 (Other: Kessler Foundation Research Center)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Disuse Osteoporosis
Keywords: Spinal Cord Injury; Disuse Osteoporosis; Zoledronic acid; Bisphosphonates; Dual Energy X-ray Absorptiometry
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zoledronic acid (Experimental): At baseline, study subjects in the treatment group will receive 5 mg of zoledronic acid (Reclast: 5 mg; Novartis Pharmaceuticals Inc., East Hanover, NJ) by intravenous infusion over 30 minutes.
  Interventions: Drug: Zoledronic acid
- No Intervention (No Intervention): Participants will receive no therapy and serve as a control group and have the same outcome measures completed at parallel time points.

INTERVENTIONS:
Drug: Zoledronic acid — At baseline, study subjects in the treatment group will receive 5 mg of zoledronic acid (Reclast: 5 mg; Novartis Pharmaceuticals Inc., East Hanover, NJ) by intravenous infusion over 30 minutes.
  Other Names: Zometa; Reclast
  Arms: Zoledronic acid

SUMMARY:
In subjects with acute SCI: To compare the effects of parenteral zoledronic acid therapy on preservation of regional and total skeletal mass (DXA).

Hypothesis: Zoledronic acid will dramatically diminish bone loss in persons with acute SCI, as evidenced by serial densitometry determinations (DXA).

DETAILED DESCRIPTION:
Immobilization is associated with disuse osteoporosis. Spinal cord injury (SCI) produces a syndrome of acute skeletal immobilization with immediate and irreversible unloading of the involved skeletal regions resulting in accelerated bone loss. In addition to rapid bone loss, there are also the complications of hypercalciuria, hypercalcemia, nephrolithiasis, and renal insufficiency. In some reports, as much as 50% of regional bone mass has been lost within the first year after paralysis. A depletion of regional bone of such magnitude greatly increases the risk of fractures, with associated morbidity and increased cost of care. Often, these fractures occur with minimal or non-obvious trauma and may pass undiagnosed for varying lengths of time due to the absence of pain sensation. The acute complications of fracture may include hemorrhage, deep venous thrombosis, and autonomic dysreflexia. Long-term complications include functional deformity, non-union, infection, heterotopic calcification, and significantly longer healing time. The sociology-economic consequences include a minimum of 1 to 2 weeks of hospitalization and the potential need for an increased level of attendant care. This study will address the efficacy of a bisphosphonate, zoledronic acid (Reclast: 5 mg; Novartis Pharmaceuticals Inc., East Hanover, NJ), in the prevention of the bone loss associated with acute SCI.

Prevention of regional osteoporosis in persons with SCI would reduce the morbidity associated with fractures, a known secondary complication of immobilization. Thus, the quality of life would be improved in terms of employment responsibilities (reduction in days absent from employment and income lost) and personal activities (recreational endeavors, independence, and ease in which one performs activities of daily living). Individuals with SCI may then engage more securely in activities without fear of fracture, a tremendous psychological benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Within 3 months of the date of acute SCI.
2. Motor-complete and incomplete SCI [American Spinal Injury Association Impairment Scale (AIS) of sensorimotor impairment (AIS A, B, and C)]

Exclusion Criteria:

1. Extensive life-threatening injuries (in addition to SCI)
2. Femur or tibia fracture or extensive bone trauma
3. History of prior bone disease (Paget's disease, overactive parathyroid, osteoporosis)
4. Post-menopausal women
5. Known allergy to bisphosphonates
6. Severe underlying chronic illness
7. Current diagnosis of cancer or history of cancer
8. I am currently receiving corticosteroids
9. Pregnancy or lactation
10. I have been diagnosed with kidney problems
11. As determined from the prescreening blood tests by the study physician Serum creatinine > 2.0 mg/dl
12. As determined from the prescreening blood tests by the study physician Corrected calcium < 8 mg/dl or > 11 mg/dl
13. As determined from the prescreening blood tests by the study physician Elevated liver function enzymes > 2 x upper limit of normal (ULN)
14. I am taking a bisphosphonate for heterotopic ossification (HO) (an overgrowth of bone typically diagnosed shortly after SCI in the pelvic region)
15. I have an existing dental condition or dental infection.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2006-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William A Bauman, M.D., Principal Investigator — James J. Peters VA Medical Center
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States

REFERENCES:
- [Background] Shapiro J, Smith B, Beck T, Ballard P, Dapthary M, BrintzenhofeSzoc K, Caminis J. Treatment with zoledronic acid ameliorates negative geometric changes in the proximal femur following acute spinal cord injury. Calcif Tissue Int. 2007 May;80(5):316-22. doi: 10.1007/s00223-007-9012-6. Epub 2007 Apr 7. PMID 17417700
- [Background] Bubbear JS, Gall A, Middleton FR, Ferguson-Pell M, Swaminathan R, Keen RW. Early treatment with zoledronic acid prevents bone loss at the hip following acute spinal cord injury. Osteoporos Int. 2011 Jan;22(1):271-9. doi: 10.1007/s00198-010-1221-6. Epub 2010 Apr 1. PMID 20358358

RESULTS

PARTICIPANT FLOW:
Groups:
- No Treatment: Participants will receive no therapy and serve as a control group and have the same outcome measures completed at parallel time points.
Period: Overall Study
Arm/Group | Zoledronic Acid | No Treatment
Started | 8 | 13
Completed | 8 | 8
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | No Treatment | Total
Number analyzed (Participants) | 8 | 13 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — Subject self reported date of birth used to calculate age
  years | 25.5 (9.6) | 33.0 (11.0) | 29.3 (20.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 12 | 19
Region of Enrollment [Number; unit: participants]
  United States | 8 | 13 | 21

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD) at the Distal Femur and Proximal Tibia at Baseline and Month 12.
Description: An imaging method known as dual energy x-ray absorptiometry (DXA) was used to obtain BMD of the distal femur and proximal tibia by using a customized research software program supplied by the manufacturer. This measurement will be the primary determinant (dependent measure) of difference among the treatment and control groups, and they will be followed over time at the previously specified time points.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Zoledronic Acid | No Treatment
Number analyzed (Participants) | 8 | 13
g/cm2
  Baseline Distal Femur | 1.102 (0.148) | 1.134 (0.244)
  12 Month Distal Femur | 0.898 (0.128) | 1.038 (0.241)
  Baseline Proximal Tibia | 1.274 (0.245) | 1.341 (1.216)
  12 Month Proximal Tibia | 1.022 (0.267) | 1.237 (0.276)

2. Secondary Outcome: Bone Mineral Density (BMD) at the Total Hip at Baseline and Month 12
Description: An imaging method known as dual energy x-ray absorptiometry (DXA) was used to obtain BMD of the total hip.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Zoledronic Acid | No Treatment
Number analyzed (Participants) | 8 | 13
g/cm2
  Baseline Total Hip | 1.125 (0.166) | 1.020 (0.154)
  12 Month Total Hip | 1.042 (0.168) | 0.814 (0.151)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Monthly assessment of medical history over the 24 month follow-up period after baseline assessment.
Arm/Group | Zoledronic Acid | No Treatment
Serious Adverse Events (participants affected / at risk) | 3/8 | 1/13
Other Adverse Events (participants affected / at risk) | 8/8 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=8) | No Treatment (N=13)
General Surgery (Surgical and medical procedures) | 3 (3) | 1 (1) — During the inpatient stay, 1 participant had gallbladder surgery, 1 participant had a suprapubic catheter inserted, 1 participant had flap surgery for a decubitus ulcer, and 1 participant had an intrathecal baclofen pump inserted.
Bowel Impaction (Gastrointestinal disorders) | 1 (1) | 0 (0) — One participant was admitted to an acute care facility for bowel impaction
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — One participant was admitted to an acute care facility for symptoms resulting from a stage IV decubitus ulcer and treatment with hyperbaric chamber therapy.
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) — Two participants were admitted to an acute care facility for sever pain that after a complete work up was diagnosed as a urinary tract infection.
Spinal headache (Nervous system disorders) | 1 (1) | 0 (0) — One participant was admitted to the hospital for severe migraine headaches. This was the result of leaking cerebral spinal fluid when spinal anesthesia punctured the dura mater during a Botulinum toxin procedure.
Deep Venous Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Patient was admitted to hospital for lower extremity pain that was diagnosed as a deep venous thrombosis.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=8) | No Treatment (N=13)
Acute Febrile Reaction (General disorders) | 6 (8) | 0 (0) — In the zoledronic acid arm, 4 participants experienced low grade fevers while 2 participants experienced moderate to severe fevers.
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0) — All subjects in the zoledronic acid arm experienced mild to severe myalgia (muscle pain).
Vomiting (Gastrointestinal disorders) | 6 (8) | 0 (0) — Vomiting was noted in 6 of the 8 participants in the zoledronic acid arm.
Lethargy (General disorders) | 8 (8) | 0 (0) — All participants in the zoledronic acid arm experienced mild to severe lethargy (drowsiness).
Hypocalcemia (Blood and lymphatic system disorders) | 1 (8) | 0 (0) — Hypocalcemia (low blood calcium) occurred in 1 participant and resolved within one week without any specific therapy instituted.

LIMITATIONS AND CAVEATS:
The clinical trial was not randomized, it had a relatively small sample size, and 5 participants received high-dose corticosteroids in an attempt to preserve neurologic function upon that could have had a profound adverse effect on the skeleton.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No